CLINICAL TRIAL: NCT07287033
Title: A Randomized, Quadruple-blinded, Placebo-controlled, Single-ascending and Multiple Dose Study to Evaluate the Safety, Local Tolerability, Pharmacokinetics, Immunogenicity, Pharmacodynamics, and Exploratory Clinical Activity of MY006 in Healthy Volunteers and Adolescent and Adult Patients With Peanut Allergy
Brief Title: Study to Evaluate the Safety, Pharmacokinetic, and Pharmacodynamic Effects of MY006 in Healthy Volunteers and Patients With Peanut Allergy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mabylon AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MY-CLN-SP-006-PA1001
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Peanut Allergies
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A, Single Ascending Dose, Dose Level 1 (Healthy Volunteers) (Experimental): Cohort A1: MY006 or Placebo, subcutaneous, single dose in healthy volunteers.
  The cohort will consist of 8 subjects. The subjects will be randomized in a 6:2 ratio in a quadruple-blinded manner to receive MY006 or Placebo (vehicle), respectively.
  Interventions: Drug: MY006 Low Dose; Drug: Placebo (Vehicle)
- Part A, Single Ascending Dose, Dose Level 2 (Healthy Volunteers) (Experimental): Cohort A2: MY006 or Placebo, subcutaneous, single dose in healthy volunteers.
  The cohort will consist of 8 subjects. The subjects will be randomized in a 6:2 ratio in a quadruple-blinded manner to receive MY006 or Placebo (vehicle), respectively.
  Interventions: Drug: MY006 Mid Dose; Drug: Placebo (Vehicle)
- Part A, Single Ascending Dose, Dose Level 3 (Healthy Volunteers) (Experimental): Cohort A3: MY006 or Placebo, subcutaneous, single dose in healthy volunteers.
  The cohort will consist of 8 subjects. The subjects will be randomized in a 6:2 ratio in a quadruple-blinded manner to receive MY006 or Placebo (vehicle), respectively.
  Interventions: Drug: MY006 High Dose; Drug: Placebo (Vehicle)
- Part A, Multiple Dose (Healthy Volunteers) (Experimental): Cohort A4: MY006 or Placebo, subcutaneous, every 2 weeks, total of 2 doses in healthy volunteers.
  The cohort will consist of 8 subjects. The subjects will be randomized in a 6:2 ratio in a quadruple-blinded manner to receive MY006 or Placebo (vehicle), respectively.
  Interventions: Drug: MY006 Selected Dose; Drug: Placebo (Vehicle)
- Part B, Single Dose with Early Peanut Challenge (Peanut-Allergic Patients) (Experimental): Cohort B1: MY006 or Placebo, subcutaneous, single dose in adults and adolescents. Peanut challenge will occur early after dosing.
  The cohort will consist of 8 subjects. The subjects will be randomized in a 6:2 ratio in a quadruple-blinded manner to receive MY006 or Placebo (vehicle), respectively.
  Interventions: Drug: MY006 Selected Dose; Drug: Placebo (Vehicle)
- Part B, Single Dose with Late Peanut Challenges (Peanut-Allergic Patients) (Experimental): Cohort B2: MY006 or Placebo, subcutaneous, single dose in adults and adolescents. Peanut challenge will occur late after dosing.
  The cohort will consist of 8 subjects. The subjects will be randomized in a 6:2 ratio in a quadruple-blinded manner to receive MY006 or Placebo (vehicle), respectively.
  Interventions: Drug: MY006 Selected Dose; Drug: Placebo (Vehicle)

INTERVENTIONS:
Drug: MY006 Low Dose — MY006 administered by subcutaneous injection.
  Arms: Part A, Single Ascending Dose, Dose Level 1 (Healthy Volunteers)
Drug: MY006 Mid Dose — MY006 administered by subcutaneous injection.
  Arms: Part A, Single Ascending Dose, Dose Level 2 (Healthy Volunteers)
Drug: MY006 High Dose — MY006 administered by subcutaneous injection.
  Arms: Part A, Single Ascending Dose, Dose Level 3 (Healthy Volunteers)
Drug: MY006 Selected Dose — MY006 administered by subcutaneous injection.
  Arms: Part A, Multiple Dose (Healthy Volunteers); Part B, Single Dose with Early Peanut Challenge (Peanut-Allergic Patients); Part B, Single Dose with Late Peanut Challenges (Peanut-Allergic Patients)
Drug: Placebo (Vehicle) — Placebo (vehicle) administered by subcutaneous injection.

SUMMARY:
The goal of this clinical trial is to evaluate the safety, pharmacokinetics, and effectiveness of MY006, a therapy designed to prevent severe or potentially life-threatening allergic reactions caused by accidental peanut intake. In the first part of the study, adult participants receive one dose or two doses of MY006 or a placebo, administered by subcutaneous injection. The safety of MY006, including the number of adverse events, injection-site reactions, and immunogenicity, in these participants will be reviewed by an independent Safety Monitoring Committee and, if the safety is judged acceptable, the second part of the study will be started. In the second part of the study, adult and adolescent participants with peanut allergy receive one dose of MY006 or a placebo, administered by subcutaneous injection. Several weeks later, the participants are given a food peanut challenge to assess reactions and treatment effects. The duration of the study for participants is for up to 32 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

Part A - Single-ascending dose and multiple dose cohorts in healthy volunteers

1. Subject is male or female between 18 to 55 years of age, inclusive, at the screening visit.
2. Subject agrees voluntarily to participate, and is able to read and understand, and willing to sign, the Institutional Review Board/Independent Ethics Committee-approved informed consent form prior to performing any screening visit procedures.
3. Subject weight at screening and admission is between 45 kg and 100 kg, inclusive.
4. Subject has a body mass index between 18.0 and 30.0 kg/m2, inclusive, at screening visit.

Part B - Peanut-allergic patient cohorts

1. Participant and/or parent/legal guardian must be able to understand and provide informed consent and/or assent, as applicable.
2. Patient is male or female between 12 to 55 years of age, inclusive, at the screening visit.
3. Patient weight at screening and admission is between 40 kg and 100 kg, inclusive.
4. If patient is 12-17 years of age, their body mass index (BMI) must be above the 5th percentile and below the 95th percentile for age and sex at the screening visit. If patient is 18 years of age or above, their BMI must be between 18.0 and 30.0 kg/m2, inclusive, at the screening visit.
5. Patient has a history of allergy to peanut and meets all of the following criteria:

   1. Positive skin prick test (≥5 mm wheal greater than Placebo) to peanut; and
   2. Positive specific IgE (≥0.7 kUA/L) to peanut and Ara h 2 at screening determined by ImmunoCap; and
   3. Positive double-blinded challenge to peanut during the screening period, defined as experiencing dose-limiting symptoms at a single dose of ≤300 mg of peanut protein.
6. Patient is willing and able to avoid peanut-containing products and any other allergy-inducing foods known to the patient for the duration of study participation.

Key Exclusion Criteria:

Part A - Single-ascending dose and multiple dose cohorts in healthy volunteers

1. Subject has a clinically relevant history, as determined by the Principal Investigator or designee, or presence of respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, and/or connective tissue diseases or disorders.
2. Subject has clinically significant abnormal vital signs, after 5 minutes or more of sitting rest, defined as any of the following:

   1. Systolic blood pressure ≥140 mmHg;
   2. Diastolic blood pressure ≥90 mmHg; and/or
   3. Heart rate ≥90 beats per minute.
3. Subject has any clinically significant abnormalities in rhythm, conduction, or morphology of the resting electrocardiogram (ECG) and/or any clinically significant abnormalities in the 12-lead ECG as considered by the Principal Investigator or designee that may interfere with the interpretation of QTc interval changes.
4. Subject has history of severe allergy/hypersensitivity, ongoing clinically significant allergy/hypersensitivity, as judged by the Principal Investigator or designee, known or suspected allergy to peanuts, and/or history of hypersensitivity to drugs with a similar structure or class.

Part B - Peanut-allergy patient cohorts

1. Patient has history of frequent or recent severe, life-threatening episodes of anaphylaxis or anaphylactic shock to peanut, as defined by more than 3 episodes of anaphylaxis within the past year and/or an episode of anaphylaxis within 60 days of screening.
2. Patient has uncontrolled or severe asthma/wheezing at screening, defined by one or more of the following criteria:

   1. Global Initiative for Asthma criteria regarding asthma control per latest guidelines;
   2. History of two or more systemic corticosteroid courses within 6 months of screening or one course of systemic corticosteroids within three months of screening to treat asthma/wheezing;
   3. Prior intubation/mechanical ventilation for asthma/wheezing;
   4. One hospitalization or emergency department visit for asthma/wheezing within 12 months of screening;
   5. Inhaled corticosteroid (ICS) dosing of >500 mcg daily fluticasone (or equivalent ICS based on the CoFAR Inhaled Corticosteroid Equivalency Tables); and/or
   6. Forced expiratory volume in one second (FEV1) <80% of predicted or FEV1/forced vital capacity <75%, with or without controller medications.
3. Patient has unstable exacerbated atopic disease (e.g., atopic dermatitis, urticaria, allergic rhinitis) defined by an episode of disease requiring initiation of systemic immunosuppressive or immunomodulatory treatment in the last 3 months.
4. Patient has current clinically significant cardiovascular, respiratory, neurologic, hepatic, hematopoietic, renal, gastrointestinal, or metabolic dysfunction unless currently controlled and stable as judged by the Principal Investigator.
5. Patient has abnormal vital signs, after 5 minutes or more of sitting rest, defined as any of the following:

   1. Systolic blood pressure ≥140 mmHg;
   2. Diastolic blood pressure ≥90 mmHg; and/or
   3. Heart rate ≥90 beats per minute.

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-06 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of Subjects with Adverse Events and Serious Adverse Events (Safety and Local Tolerability) | From dosing (Day 1) to End of Study visit (Part A, Week 24 or 26; Part B, Week 24/25)
  The nature of the adverse event (AE), date of the AE onset, date of the AE outcome to date, severity of the AE, and action taken for the AE will be documented together with the Principal Investigator's assessment of the seriousness of the AE and causal relationship to study drug and/or study procedure. The AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 21.0 or higher.

SECONDARY OUTCOMES:
Pharmacokinetics: Cmax (Part A, Cohorts A1-A4; Part B, Cohorts B1-B2) | From dosing (Day 1) to End of Study visit (Part A, Week 24 or 26; Part B, Week 24/25)
  Maximum serum MY006 concentration in cohorts of adult healthy volunteers (Part A) and peanut-allergic patients (Part B)
Pharmacokinetics: Tmax (Part A, Cohorts A1-A4; Part B, Cohorts B1-B2) | From dosing (Day 1) to End of Study visit (Part A, Week 24 or 26; Part B, Week 24/25)
  Time to reach Cmax of MY006 in cohorts of adult healthy volunteers (Part A) and peanut-allergic patients (Part B)
Pharmacokinetics: AUClast (Part A, SAD, Cohorts A1-A3) | From dosing (Day 1) to End of Study visit (Week 24)
  Area under the concentration-time curve (AUC) from Pre-Dose (time 0) to the time of the last quantifiable concentration (tlast) in single ascending dose (SAD) cohorts of adult healthy volunteers (Part A)
Pharmacokinetics: AUClast (Part A, MD, Cohort A4) | From Day 15 to End of Study visit (Week 26)
  AUC from Pre-Dose on Day 15 (time 0) to the time of the last quantifiable concentration (tlast) following last dose in multiple dose (MD) cohort of adult healthy volunteers (Part A)
Pharmacokinetics: AUC0-504hr (Part A, SAD, Cohorts A1-A3) | From dosing (Day 1) to Day 21
  AUC from Pre-Dose (time 0) to 504 hours post-dosing in single ascending dose (SAD) cohorts of adult healthy volunteers (Part A)
Pharmacokinetics: AUC0-336hr (Part B, Cohorts B1-B2) | From dosing (Day 1) to Day 14
  AUC from Pre-Dose (time 0) to 336 hours postdosing in peanut-allergic patients (Part B)
Pharmacokinetics: AUC0-336hr (Part A, MD, Cohort A4) | From dosing (Day 1) to Day 14
  AUC from Pre-Dose (time 0) to 336 hours post-dosing in multiple dose (MD) cohort of adult healthy volunteers (Part A)
Pharmacokinetics: AUCinf (Part A, SAD, Cohorts A1-A3; Part B, Cohorts B1-B2) | From dosing (Day 1) to End of Study visit (Week 24/25)
  AUC from Pre-Dose (time 0) extrapolated to infinite time in single ascending dose (SAD) cohorts of adult healthy volunteers (Part A) and peanut-allergic patients (Part B)
Pharmacokinetics: AUCinf (Part A, MD, Cohort A4) | From Day 15 to End of Study visit (Week 26)
  AUC from Pre-Dose on Day 15 (time 0) extrapolated to infinite time in multiple dose (MD) cohort of adult healthy volunteers (Part A)
Pharmacokinetics: AUC%extrap (Part A, Cohorts A1-A4; Part B, Cohorts B1-B2) | From dosing (Day 1) to End of Study visit (Part A, Week 24 or Week 26; Part B, Week 24/25)
  Percentage of AUCinf that is due to extrapolation beyond tlast in cohorts of adult healthy volunteers (Part A) and peanut-allergic patients (Part B)
Pharmacokinetics: λz (Part A, MD, Cohort A4; Part B, Cohorts B1-B2) | From dosing (Day 1) to End of Study visit (Week 24/25)
  Terminal elimination rate constant in multiple dose (MD) cohort of adult healthy volunteers (Part A) and peanut-allergic patients (Part B)
Pharmacokinetics: t½ (Part A, MD, Cohort A4; Part B, Cohorts B1-B2) | From dosing (Day 1) to End of Study visit (Part A, Week 26; Part B, Week 24/25)
  Terminal elimination half-life in multiple dose (MD) cohort of adult healthy volunteers (Part A) and peanut-allergic patients (Part B)
Pharmacokinetics: CL/F (Part A, MD; Cohort A4, Day 15; Part B, Cohorts B1-B2) | From dosing (Day 1) to Day 15 (Part A) or End of Study visit (Part B, Week 24/25)
  Total body clearance in multiple dose (MD) cohort of adult healthy volunteers (Part A) and peanut-allergic patients (Part B)
Pharmacokinetics: Vz/F (Part A, MD, Cohort A4, Day 15; Part B, Cohorts B1-B2) | From dosing (Day 1) to End of Study visit (Part A, Week 26; Part B, Week 24/25)
  Apparent volume of distribution in multiple dose (MD) cohort of adult healthy volunteers (Part A) and peanut-allergic patients (Part B)
Pharmacokinetics: Racc,Cmax (Part A, MD, Cohort A4) | From dosing (Day 1) to Day 15
  Ratio of last dose Cmax (Day 15) to first dose Cmax (Day 1) in multiple dose (MD) cohort of adult healthy volunteers (Part A)
Pharmacokinetics: Racc,C72 (Part A; MD; Cohort A4) | From dosing (Day 1) to Day 18
  Ratio of MY006 concentration at 72 hours (C72) post Day 15 to first dose C72 (Day 1) in multiple dose (MD) cohort of adult healthy volunteers (Part A)
Pharmacokinetics: Racc,C168 (Part A, MD, Cohort A4) | From Day 8 to Day 22
  Ratio of MY006 concentration at 168 hours (C168) post Day 15 dose to first dose C168 (Day 1) in multiple dose (MD) cohort of adult healthy volunteers (Part A)
Pharmacokinetics: Racc,AUC0-336hr (Part A, MD, Cohort A4) | From dosing (Day 1) to Day 15
  Ratio of last dose AUC0-336hr (Day 15) to first dose AUC0-336hr (Day 1) in multiple dose (MD) cohort of adult healthy volunteers (Part A)
Immunogenicity: ADA (Part A, Cohorts A1-A4; Part B, Cohorts B1-B2) | From dosing (Day 1) to End of Study visit (Part A, Week 24 or 26; Part B, Week 24/25)
  Percentage of subjects developing treatment-emergent anti-drug antibodies (ADA)
Immunogenicity: Treatment-enhanced ADA (Part A, Cohorts A1-A4; Part B, Cohorts B1-B2) | From dosing (Day 1) to End of Study visit (Part A, Week 24 or 26; Part B, Week 24/25)
  Percentage of subjects developing treatment-enhanced ADA
Immunogenicity: ADA Titers (Part A, Cohorts A1-A4; Part B, Cohorts B1-B2) | From dosing (Day 1) to End of Study visit (Part A, Week 24 or 26; Part B, Week 24/25)
  Amount of ADA in subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Syneos Health Clinical Research Services LLC, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No